CLINICAL TRIAL: NCT04321863
Title: Stratifying Crohn's Using Biomarker Assessment
Acronym: SCUBA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: 20/WS/0028; 246230 (Other: IRAS ID)
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Crohn Disease in Remission
Keywords: Faecal biomarkers; Serum biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with Crohn's disease in remission: All patients recruited will submit two samples to facilitate faecal zinc and qFIT in addition to FC which is standard of care. All patients recruited will have an additional tube of blood taken to measure serum zinc at the same time as they have their routine (standard of care) monitoring bloods taken - no additional venepuncture will be required.
  Interventions: Other: Faecal calprotectin (FC); Other: quantitative Faecal Immunochemical Testing (qFIT); Other: Serum and faecal zinc

INTERVENTIONS:
Other: Faecal calprotectin (FC) — FC is a surrogate marker of neutrophil influx into the gut lumen. It accurately predicts mucosal healing (MH) at colonoscopy, and thus is already widely used in clinical practice in disease monitoring in CD patients (standard of care).
Other: quantitative Faecal Immunochemical Testing (qFIT) — Stool test for haemoglobin. It has been shown to predict mucosal healing in Crohn's disease and ulcerative colitis. This study will compare the ability of qFIT and FC to predict flare in CD (qFIT is a cheaper, more stable test with a quicker turn-around time than FC, and is also less labour intensive for the lab).
Other: Serum and faecal zinc — Blood sample for serum zinc will be taken at same time as routine (standard of care) monitoring bloods which include CRP - no additional venipuncture will be required. A single stool sample will be sufficient to measure FC (as outlines above) and faecal zinc. This study will compare the ability of serum/faecal zinc and CRP at predicting relapse in patients with quiescent (inactive) luminal (affecting the small and/or large bowel) CD.

SUMMARY:
Crohn's disease (CD) is a relapsing-remitting condition that requires lifelong monitoring. Non-invasive tests such as faecal calprotectin (FC) are more acceptable to patients and cost-effective than invasive tests such as colonoscopy.

FC levels can also accurately predict the degree of healing seen within the bowel at colonoscopy.

FC testing is labour intensive, and results are often indeterminate. There is interest in a newer test called quantitative Faecal Immunochemical Testing (qFIT) in patients with CD. qFIT measures the amount of blood within the stool and is used in the Scottish Bowel Cancer Screening Programme. qFIT is an easier and more acceptable test for patients and is less labour intensive and cheaper for the lab to process than FC.

qFIT is a useful test to 'rule-out' significant colorectal pathology including bowel cancer, high risk polyps and inflammatory bowel disease in patients in the primary care setting. It has also been used to predict the degree of healing seen within the bowel at colonoscopy and to predict the risk of relapse in patients with UC, but not in CD. There are no studies in the UK to date comparing FIT to FC as a monitoring test in patients with well-controlled CD.

Unpublished audit data from our group has suggested that low serum zinc has higher predictive accuracy at determining risk of future flare than both FC and CRP; we are unsure if this is due to higher faecal losses in 'grumbling' CD patients.

This study could identify a cheaper, more acceptable and easier to interpret test to guide disease activity monitoring, flare risk and treatment decisions in quiescent CD.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a relapsing and remitting condition requiring lifelong monitoring.

Stool sampling for disease monitoring in inflammatory bowel disease (IBD) is non-invasive, cost-effective and acceptable to patients. Faecal calprotectin (FC) and quantitative Faecal Immunochemical Testing (qFIT) are both stool-based tests.

FC is a surrogate marker of neutrophil influx into the gut lumen. It accurately predicts mucosal healing (MH) at colonoscopy, and thus FC is already widely used in clinical practice in disease monitoring in CD patients.

qFIT, testing stool for haemoglobin, has been used in the Scottish Bowel Cancer Screening Programme since November 2017. A 'negative' qFIT is also a useful 'rule-out' test for significant colorectal pathology (including colorectal cancer, high-risk adenomas and IBD) in primary care. qFIT has been shown to predict MH in both CD and ulcerative colitis (UC), and has been used to predict relapse in patients with UC but not CD. There is no UK study to date comparing the ability of qFIT and FC to predict flare in CD.

qFIT is a cheaper, more stable test with a quicker turn-around time than FC. It is also less labour intensive for the lab.

CRP is a cheap and easily available biomarker but is insensitive, non-specific and inferior to FC at predicting relapse in CD. CRP can also be elevated by infective complications or other concomitant inflammatory disease which makes its interpretation difficult. New data from our group has suggested that low serum zinc has higher predictive accuracy at determining risk of future flare than both FC and CRP; we are unsure if this is due to higher faecal losses in 'grumbling' CD patients.

This observational, prospective cohort study will recruit patients with luminal (affecting small and/or large bowel) CD in clinical remission (i.e. asymptomatic). A stool sample will be used to check a qFIT and faecal zinc in addition to the routinely monitored FC. At the time of routine blood collection, an additional sample will be taken to check plasma zinc. CRP is already checked routinely.

Patients will be followed up for one year, or until flare/relapse - this information will be accessed remotely through electronic patient records.

The ability of qFIT, serum zinc and faecal zinc to predict relapse in CD will be compared to FC using area under the ROC curve (AUC).

Primary study aim:

To compare the ability of qFIT and FC at predicting relapse/flare in patients with quiescent (inactive) luminal (affecting the small and large bowel) CD.

Relapse (or flare) is defined as the need for new or additional treatment for CD, hospitalisation for CD, or CD related surgery.

Primary hypothesis:

qFIT is not inferior to FC at predicting flare in quiescent (inactive) luminal (affecting the small and large bowel) CD.

Secondary study aim:

Compare the ability of serum/faecal zinc and CRP at predicting relapse in patients with quiescent (inactive) luminal (affecting the small and/or large bowel) CD.

Secondary hypothesis:

Serum/faecal zinc is superior to CRP at predicting relapse/flare in patients with quiescent (inactive) luminal (affecting the small and large bowel) CD.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of luminal CD by standard endoscopic, histological or radiological criteria
2. In clinical remission as defined by Harvey Bradshaw Index (HBI) <4
3. Aged 18-50
4. On any CD-related therapy or indeed no therapy
5. Having FC checked anyway to monitor mucosal disease activity

Exclusion Criteria:

1. Isolated perianal or upper GI CD
2. Short gut syndrome necessitating total parenteral nutrition (TPN); otherwise patients with stomas allowed.
3. Current or previous colorectal carcinoma or high-risk adenoma, active diverticular disease (diverticulitis) or haemorrhoids
4. Ulcerative or indeterminate colitis
5. Patients taking NSAIDs, warfarin, heparin, anti-platelet therapy or DOACs.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with quiescent (inactive) luminal Crohn's disease attending secondary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Estimated)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
qFIT and FC | 1 year
  To compare the ability of qFIT and FC at predicting relapse/flare in patients with quiescent (inactive) luminal (affecting the small and large bowel) CD.
  Relapse (or flare) is defined as the need for new or additional treatment for CD, hospitalisation for CD, or CD related surgery.
  The ability of qFIT to predict relapse in CD will be compared to FC using area under the ROC curve (AUC).

SECONDARY OUTCOMES:
Serum/faecal zinc | 1 year
  Compare the ability of serum/faecal zinc and CRP at predicting relapse in patients with quiescent (inactive) luminal (affecting the small and/or large bowel) CD. Relapse (or flare) is defined as the need for new or additional treatment for CD, hospitalisation for CD, or CD related surgery.
  The ability of serum zinc and faecal zinc to predict relapse in CD will be compared to FC using area under the ROC curve (AUC).

CONTACTS AND LOCATIONS:
Locations (1):
- Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No